CLINICAL TRIAL: NCT03846726
Title: Watch-and-wait Approach Versus Surgical Resection for Rectal Cancer Patients With Complete Clinical Response After Chemoradiotherapy: a Multi-center Cohort Study
Brief Title: Treatment Strategy for Rectal Cancer Patients With Complete Clinical Response
Status: Completed | Type: Observational
Sponsor: Yuan-hong Gao (Other)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other); Peking University Cancer Hospital & Institute (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Fujian Medical University Union Hospital (Other); Fujian Cancer Hospital (Other Government); Tongji Hospital (Other)
Responsible Party: Sponsor-Investigator, Yuan-hong Gao, Principal Investigator, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: B2018-174-01
Record Dates: First submitted 2019-01-22; First posted 2019-02-20 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Rectal Cancer; Organ Preservation
Keywords: Rectal Cancer; clinical complete response
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- observation group: Pathologically confirmed stage II/III rectal adenocarcinoma patients who received neoadjuvant chemoradiotherapy followed by a clinical complete response, and refused surgery but went on with the watch and wait approach.
- surgery group: Pathologically confirmed stage II/III rectal adenocarcinoma patients who received neoadjuvant chemoradiotherapy followed by a clinical complete response, and received radical resection.
  Interventions: Procedure: standard TME surgery

INTERVENTIONS:
Procedure: standard TME surgery — radical resection for rectal cancer
  Groups: surgery group

SUMMARY:
This was a propensity-score matched observational analysis, comparing the oncological outcome of surgical resection vs watch and wait apporach for rectal cancer patients with a cCR.

DETAILED DESCRIPTION:
Pathologically confirmed stage II/III rectal adenocarcinoma patients who received neoadjuvant chemoradiotherapy followed by a clinical complete response from the year 2010 to 2018 were included. Sequential subjects were identified from a prospective maintained database in the Sun Yat-sen University Cancer Center. Clinical experts on rectal cancer from other 5 regional medical centers in China were also invited to participate, and provided data of cCR patients. Standardized forms for data collection were sanded to researchers in each center. Patients received radical resection will constituted our surgery group. Those refused surgery constituted the observation group who went on with the watch and wait approach. A propensity-score matched observational analysis will be used to compare the oncological outcome of these two groups.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed stage II/III rectal adenocarcinoma patients who received neoadjuvant chemoradiotherapy followed by a clinical complete response

Exclusion Criteria:

* history of a second primary malignancy.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pathologically confirmed stage II/III rectal adenocarcinoma patients who received neoadjuvant chemoradiotherapy followed by a clinical complete response were included and divided into two groups according to the treatment followed.
Sampling Method: Non-Probability Sample
Enrollment: 513 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
PFS | the time from the date of treatment started until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  progression-free survival

SECONDARY OUTCOMES:
OS | Overall survival was calculated from the date of first treatment until death from any cause or was censored at last follow-up, assessed up to 60 months
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-hong Gao, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided